CLINICAL TRIAL: NCT02158897
Title: Effect of a Periodic Fasting-mimicking Diet on Risk Factors for Metabolic Syndrome and Age-related Diseases
Brief Title: Multi-cycle Prolon Diet
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Min Wei, Research assistant professor, University of Southern California
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HS-12-00391
Record Dates: First submitted 2014-06-02; First posted 2014-06-09 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Control (No Intervention): Participants will consume their normal diet. Body weight and physiological change at two time points (approximately 2-3 months apart) will be examined. The participants will be crossed over to the diet group.
- Prolon Diet (Experimental): Participants will be provided with a 5-day supply of fasting-mimicking diet, including energy bars, soups, drink packets and dietary supplements. Participants will diet for 3 cycles. Each one-month cycle consists of 5 days of dieting with a calorie intake estimated at 600-1200 calories per day. The rest of the month participants will eat normally. After 3 cycles, participants will be examined again after consuming their normal diet after 2-3 months.
  Interventions: Other: Prolon diet

INTERVENTIONS:
Other: Prolon diet — 3 cycles of a 5-day Prolon diet very month
  Other Names: Fasting-mimicking diet
  Arms: Prolon Diet

SUMMARY:
Evidence from bio-gerontology research from our laboratory and others have showed that short-term fasting/starvation (STS) can improve the efficacy of chemotherapy by protecting normal cells and tissues and potentially sensitizing malignant cells to chemo drugs. Furthermore, STS improves risk factors associated with aging and age-related disease in rodent models. Prolonged fasting, however, is difficult to implement and may not be feasible or safe in humans. We have developed a fasting-mimicking diet (FMD) that was well accepted in a pilot human trial. The objective of the study is to ascertain the impact of the fasting-mimicking diet given to adult subjects for 5 days a month for 3 consecutive months. The investigators hypothesize that the specially designed dietary regimen can reduce the risk factors for metabolic syndrome and biomarkers associated with aging and age-related diseases.

DETAILED DESCRIPTION:
The Phase I part of the study is designed as a randomized cross-over trial, including two arms: a Control arm and a multi-cycle special 5-day dietary regimen (Diet, 3 cycles) arm. After 3 cycles, the Control and Diet groups are crossed over such that the Control group will under-go dieting and the Diet group will return to normal diet. Participants will be monitored for body weight and physiological changes, as well as the adherence to the dietary intervention.

The Phase II part of the study is an expansion of the Phase I to ascertain the impact of the dietary intervention on risk factors for metabolic syndrome and biomarkers associated with aging and age-related diseases.

Statistical methods: Paired samples t-test and Mann-Whitney test will be used to compare between Control and Diet groups as well as pre- and post-diet values.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy adults
* BMI >19 kg/m^2

Exclusion Criteria:

* Severe hypertension (systolic BP > 200 mm Hg and/or diastolic BP > 105 mm Hg).
* Underweight (BMI < 19 kg/m^2)
* Females who are pregnant or nursing
* Special dietary requirements incompatible with the study interventions
* Significant food allergies which would make the subject unable to consume the study food
* Alcohol dependency (alcohol intake greater than two drinks per day for women and three drinks per day for men).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2013-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Safety and feasibility of the Prolon diet | 1 and half years
  Phase I: To obtain preliminary estimates of the feasibility and safety of a low calorie Prolon diet in adult subjects.
Effect of Prolon diet on risk factors for metabolic syndrome and biomarkers of aging | 2 and half years
  Phase II: To ascertain the impact of the calorie restricted special diet on the risk factors for metabolic syndrome and biomarkers associated with aging and age-related diseases: e.g. fasting glucose, glucose tolerance, blood pressure, abdominal obesity, lipid profile, circulating IGF-1 and IGFBP1.

SECONDARY OUTCOMES:
Changes in cognitive functions before and after the dietary intervention. | 2 and half years
  Effects of dieting on the brain using fMRI;
  Effects of dieting on cognitive functions:
  1. Verbal memory and learning;
  2. Speed of processing/attention;
  3. Working memory;
  4. Executive function;
  5. Visuospatial construction and memory;
  6. Frequency of Forgetting;

CONTACTS AND LOCATIONS:
Locations (1):
- Davis School of Gerontology, Los Angeles, California, United States